CLINICAL TRIAL: NCT06756529
Title: The Effect of Hand Massage on Pain, Anxiety, Fear and Nausea After Surgery in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Akıl (Other)
Responsible Party: Sponsor-Investigator, Fatma Akıl, principal investigator, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fatma
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Hand Massage; Pain; Anxiety; Fear; Nausea-vomiting; Child; Nurse
Keywords: hand massage; pain; anxiety; fear; nausea-vomiting; child; nurse
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): group receiving hand massage
  Interventions: Other: hand massage
- control group (No Intervention): Group without hand massage

INTERVENTIONS:
Other: hand massage — Hand massage was applied to the patients before surgery, on the morning of surgery and after surgery.
  Other Names: experimental group
  Arms: experimental group

SUMMARY:
This study was conducted to determine the effect of hand massage on postoperative anxiety, pain, fear, and nausea and vomiting after pediatric surgery. This is a randomized, controlled experimental study. The sample consisted of 107 sick children who underwent ingunial hernia surgery (control: 55; experimental: 52). Hand massage was applied to the sick children in the experimental group the day before the surgery, on the morning of the surgery and after the surgery.

DETAILED DESCRIPTION:
Due to various diseases throughout their developmental period, children find themselves in an environment where painful procedures are performed that they have not experienced before, and they remain in the hospital due to their illnesses. Surgical procedures constitute a portion of children's hospitalizations. Being exposed to unknown tools and physically painful procedures, being away from the family, and being in a foreign environment are situations that cause the child and family to experience anxiety. Children's anxieties about illness and hospital cause negative consequences such as prolonged recovery time and increased need for pain and sedative medication. Children's fears and anxieties about injuries and medical procedures reduce compliance with the treatment process and cause treatment to be delayed or postponed. Excessive anxiety hinders children's effectiveness in coping with medical treatment and increases uncooperative behavior and negative emotions toward healthcare professionals. Anxiety and pain are considered two common problems experienced by children before and after surgery. Pain causes changes in the brain and makes future pain worse. It slows healing, impairs treatment, and causes medical problems. Untreated pain causes anxiety, depression, irritability, and fatigue. Pain is a common consequence of surgery worldwide, and unrelieved or poorly managed pain is a burden on the child, the healthcare system and society.

Many patients described nausea and vomiting as the most unpleasant surgery-related experience they had in the postoperative period, even more than pain. In particular, prolonged hospital stay leads to re-admission and therefore increased treatment costs. At the same time, it causes the time allocated for nursing care to be prolonged, causing negative reflections on work-time management and therefore on the quality of patient care. Therefore, early detection and prevention of postoperative nausea and vomiting is very important for the satisfaction of the child and family and the quality of care.

In the literature, many non-pharmacological applications such as letting sick children listen to music, virtual reality glasses, and games after surgery have been performed and their effects on parameters such as pain, nausea-vomiting, and anxiety have been examined. Although there are studies examining the relationship between postoperative hand massage and anxiety, pain, fear and nausea in children, they are limited. Therefore, the aim of this study is to determine the effect of hand massage on anxiety, pain, fear and nausea and vomiting in children who have ingunial hernia surgery and are hospitalized in the pediatric surgery clinic.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 7-12,
* Pediatric patients who are scheduled for ingunial hernia surgery,
* Volunteers to participate in the research,
* Those whose families agree to participate in the research
* No communication problems (vision, hearing, mental),
* For patients in the experimental group; All patients who did not have an infectious disease on the hand skin (shingles, fungus, eczema, warts, calluses), local infection (abscess, etc.), open lesion/wound, scar tissue, edema, hematoma, recent fracture or dislocation were included in the sample.

Exclusion Criteria:

* Being outside the 7-12 age range,
* Pediatric patients for whom ingunial hernia surgery is not planned,
* Those who do not volunteer to participate in the research,
* The family does not agree to participate in the research
* Having communication problems
* For patients in the experimental group, patients with infectious diseases, lesions, open wounds, hematomas, fractures-dislocations on the skin of the hands were not included in the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale | one day before surgery
  This scale, consisting of 20 items, aims to evaluate the relationship of parameters such as tension, uneasiness, anxiety, and irritability with state anxiety. If the child indicates the presence of these parameters as 'a lot', 3 points are given, if the child indicates 'little', 2 points are given, and if the child indicates that they are not present at all, 1 point is given. The total score obtained from each scale is between 20-80.
State-Trait Anxiety Scale | the morning of surgery
  This scale, consisting of 20 items, aims to evaluate the relationship of parameters such as tension, uneasiness, anxiety, and irritability with state anxiety. If the child indicates the presence of these parameters as 'a lot', 3 points are given, if the child indicates 'little', 2 points are given, and if the child indicates that they are not present at all, 1 point is given. The total score obtained from each scale is between 20-80.
State-Trait Anxiety Scale | 1st day after surgery
  This scale, consisting of 20 items, aims to evaluate the relationship of parameters such as tension, uneasiness, anxiety, and irritability with state anxiety. If the child indicates the presence of these parameters as 'a lot', 3 points are given, if the child indicates 'little', 2 points are given, and if the child indicates that they are not present at all, 1 point is given. The total score obtained from each scale is between 20-80.
Wong Baker Pain Rating Scale | one day before surgery
  It contains a total of 6 facial expressions. Scoring is made between zero and five. "I have no pain", "I have mild pain", "I have moderate pain", "I have a lot of pain", "I have severe pain" and "I have severe pain" and "I have no pain" corresponding to each score, starting from the low score. With the expressions "I have very severe pain", the facial expression shape that is close to the patient's facial expression is determined and scoring is made according to this determined shape.
Wong Baker Pain Rating Scale | the morning of surgery
  It contains a total of 6 facial expressions. Scoring is made between zero and five. "I have no pain", "I have mild pain", "I have moderate pain", "I have a lot of pain", "I have severe pain" and "I have severe pain" and "I have no pain" corresponding to each score, starting from the low score. With the expressions "I have very severe pain", the facial expression shape that is close to the patient's facial expression is determined and scoring is made according to this determined shape.
Wong Baker Pain Rating Scale | 1st day after surgery
  It contains a total of 6 facial expressions. Scoring is made between zero and five. "I have no pain", "I have mild pain", "I have moderate pain", "I have a lot of pain", "I have severe pain" and "I have severe pain" and "I have no pain" corresponding to each score, starting from the low score. With the expressions "I have very severe pain", the facial expression shape that is close to the patient's facial expression is determined and scoring is made according to this determined shape.
Medical Fear Scale | one day before surgery
  This scale is a three-choice Likert type scale. For each question on the scale, a person is asked to choose one of the options "I am not at all afraid (1), I am a little afraid (2), I am very afraid (3) and the scale score is calculated. The lowest score on the scale is 27 and the highest score is 87. Children with a score between "0-29" are considered as less afraid, children with a score between "29-58" are considered as slightly afraid, and children with a score between "58-87" are considered as very afraid.
Medical Fear Scale | the morning of surgery
  This scale is a three-choice Likert type scale. For each question on the scale, a person is asked to choose one of the options "I am not at all afraid (1), I am a little afraid (2), I am very afraid (3) and the scale score is calculated. The lowest score on the scale is 27 and the highest score is 87. Children with a score between "0-29" are considered as less afraid, children with a score between "29-58" are considered as slightly afraid, and children with a score between "58-87" are considered as very afraid.
Medical Fear Scale | 1st day after surgery
  This scale is a three-choice Likert type scale. For each question on the scale, a person is asked to choose one of the options "I am not at all afraid (1), I am a little afraid (2), I am very afraid (3) and the scale score is calculated. The lowest score on the scale is 27 and the highest score is 87. Children with a score between "0-29" are considered as less afraid, children with a score between "29-58" are considered as slightly afraid, and children with a score between "58-87" are considered as very afraid.
Baxter Nausea Facial Expressions Scale (BARF Scale) | one day before surgery
  This scale, consisting of 6 different facial expressions, is evaluated between 0-10 points and there are two points between each facial expression.
Baxter Nausea Facial Expressions Scale (BARF Scale) | the morning of surgery
  This scale, consisting of 6 different facial expressions, is evaluated between 0-10 points and there are two points between each facial expression.
Baxter Nausea Facial Expressions Scale (BARF Scale) | 1st day after surgery
  This scale, consisting of 6 different facial expressions, is evaluated between 0-10 points and there are two points between each facial expression.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No